CLINICAL TRIAL: NCT01005069
Title: Phase-II Clinical Study: A Randomized, Double Blind, Dose Ranging, and Controlled Study to Evaluate the Efficacy of DLBS-32 in Subjects With Type-II Diabetes Mellitus
Brief Title: Efficacy of DLBS-32 in Subjects With Type-II Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS-32-0309
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; DLBS-32; fasting plasma glucose; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Treatment I (Experimental)
  Interventions: Drug: DLBS-32
- Treatment II (Experimental)
  Interventions: Drug: DLBS-32
- Treatment III (Experimental)
  Interventions: Drug: DLBS-32
- Treatment IV (Experimental)
  Interventions: Drug: DLBS-32
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: DLBS-32 — DLBS-32 50 mg once daily and lifestyle modification
  Arms: Treatment I
Drug: DLBS-32 — DLBS-32 100 mg once daily and lifestyle modification
  Arms: Treatment II
Drug: DLBS-32 — DLBS-32 200 mg once daily and lifestyle modification
  Arms: Treatment III
Drug: DLBS-32 — DLBS-32 300 mg once daily and lifestyle modification
  Arms: Treatment IV
Drug: Placebo capsule — Placebo capsules once daily and lifestyle modification
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate clinical efficacy and safety of DLBS 32 in the management of subjects with type-II-diabetes mellitus and to determine the minimal effective dose of DLBS 32 for subjects with type-II-diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Fasting capillary blood glucose of 127-249 mg/dL at screening
* BMI >= 18.5 kg/m^2 or waist circumference of >= 90 cm (male) or >= 80 cm (female)
* Normal liver function
* Normal renal function
* OHA-naive type-II-diabetic patients

Exclusion Criteria:

* Symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Uncontrolled hypertension
* History of or current treatment with insulin
* Current treatment with systemic corticosteroids or herbal (alternative) medicines
* History of renal and/or liver disease
* Pregnant or breast feeding females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction of venous Fasting Plasma Glucose from baseline | every 2-week interval over 6 weeks of treatment

SECONDARY OUTCOMES:
Reduction of 2h-post-prandial plasma glucose from baseline | six weeks
Change of homeostasis model assessment of insulin resistance (HOMA-IR) from baseline | six weeks
Change of high sensitivity C-reactive protein (hs-CRP) from baseline | six weeks
Liver Function, Renal Function, Adverse events | six weeks
Change in HbA1c from baseline | six weeks
Change in lipid profile from baseline | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ketut Suastika, Prof. Dr., Principal Investigator — Division of Endocrinology and Metabolic Disease University of Udayana / Sanglah Denpasar Hospital; Nuniek E Nugrahini, Dr., Principal Investigator — Department of internal medicine, RSUD Tarakan
Locations (2):
- Indonesia (2):
  - Sanglah Hospital Denpasar, Denpasar, Bali
  - RSUD Tarakan, Jakarta Pusat, DKI Jakarta